CLINICAL TRIAL: NCT02406833
Title: A Phase I, Open-Label, Dose-Escalation Study to Investigate the Safety of ISTH0036, a 'Next Generation' TGF-β2-Selective Antisense Oligonucleotide, in Subjects With Primary Open-Angle Glaucoma Undergoing Trabeculectomy
Brief Title: Phase I Dose Escalation Study to Investigate the Safety of ISTH0036 in Subjects With Glaucoma Undergoing Trabeculectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Isarna Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISTH-01-111; 2014-004985-74 (EudraCT Number)
Record Dates: First submitted 2015-03-25; First posted 2015-04-02 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Primary Open Angle Glaucoma
Keywords: glaucoma; trabeculectomy
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — ISTH0036; Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TGF-β2 antisense oligonucleotide (Experimental): Core Study: Administered intravitreally at the time of trabeculectomy at escalating doses
  Post-Study Follow-up: until 1 year after administration
  Interventions: Drug: TGF-β2 antisense oligonucleotide; Procedure: Trabeculectomy

INTERVENTIONS:
Drug: TGF-β2 antisense oligonucleotide — intravitreal injection
  Other Names: ISTH0036
Procedure: Trabeculectomy — Standard trabeculectomy with the use of antimetabolites (mitomycin C) for glaucoma patients with insufficient intraocular pressure (IOP) control

SUMMARY:
This study evaluates the addition of ISTH0036, an antisense oligonucleotide against TGF-β2, to glaucoma filtration surgery (trabeculectomy). The treatment aims at improving the surgery outcome by prevention of excessive scarring and trabecular meshwork transformation.

DETAILED DESCRIPTION:
The transforming growth factor beta (TGF-β) is known to play a key role in glaucoma. Increased levels of TGF-β2 in the eye have been linked to trabecular meshwork transformation, increased intraocular pressure and direct optic nerve damage.

Trabeculectomy is the standard surgical intervention to reduce intraocular pressure in subjects no longer sufficiently responding to pressure-lowering medications. Scarring of the surgically opened canal (bleb) often abolishes the effect of trabeculectomy (despite the intraoperative use of Mitomycin C to prevent this). TGF-β2 has been described to play a distinct role in the fibrotic process of bleb closure.

ELIGIBILITY:
Inclusion Criteria:

* Subject scheduled for trabeculectomy with Mitomycin C
* Subject no longer tolerating or benefitting from pharmacologic treatment of glaucoma

Exclusion Criteria:

* History of relevant ocular trauma < 6 months or ocular infection/inflammation < 3 months
* severe central visual field loss within 6 months unrelated to glaucoma
* pregnant or nursing women or subjects not using adequate contraception
* history or evidence of any other clinically significant disorder, condition or disease that would pose a risk to subject safety or interfere with study evaluations, procedures or interpretation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by clinical monitoring and reporting of adverse events (AE) and serious adverse events (SAE) | 1 year

SECONDARY OUTCOMES:
Intraocular pressure | 1 year
Number of interventions post trabeculectomy | 1 year
Visual field | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Petra Fettes, PhD, Study Director — Isarna Therapeutics
Locations (3):
- Germany (3):
  - University Hospital Magdeburg, Ophthalmology, Magdeburg
  - Department of Ophthalmology, Johannes-Gutenberg University Mainz, Mainz
  - University of Tuebingen, Center of Ophthalmology, Tübingen